CLINICAL TRIAL: NCT02996890
Title: Double Blinded, Randomized, Placebo Controlled, Dose Finding Trial to Evaluate the Optimal Dose of MV-ZIKA, a New Vaccine Against Zika Virus, in Regard to Immunogenicity, Safety, and Tolerability in Healthy Volunteers
Brief Title: Zika-Vaccine Dose Finding Study Regarding Safety, Immunogenicity and Tolerability (V186-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V186-001; 2016-004212-34 (EudraCT Number); MV-ZIKA-101 (Other: Themisbio)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Zika Virus
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose - single shot (Experimental): MV-ZIKA, high dose, one vaccination, day 0
  Interventions: Biological: MV-ZIKA; Other: Placebo
- Low dose (Experimental): MV-ZIKA, low dose, two vaccinations, day 0 and day 28
  Interventions: Biological: MV-ZIKA
- High dose (Experimental): MV-ZIKA, high dose, two vaccinations, day 0 and day 28
  Interventions: Biological: MV-ZIKA
- Placebo (Placebo Comparator): Physiological saline, two treatments
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MV-ZIKA — MV-Zika vaccine
  Arms: High dose; High dose - single shot; Low dose
Other: Placebo — physiological saline
  Arms: High dose - single shot; Placebo

SUMMARY:
Double blinded, randomized, placebo-controlled, dose finding, multi-center, phase 1 trial in 48 healthy volunteer subjects.

After completion of screening procedures, the subjects are randomized to one of four treatment groups (different dosage strengths and placebo) All subjects will receive study treatment at day 0 and will return on day 28. Subjects randomized to treatment groups with two vaccinations will receive a second treatment at day 28.

Subjects will return on day 56 for the final visit.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers aged 18 to 55
* subjects of child bearing potential must perform reliable method of contraception

Exclusion Criteria:

* immune deficiency, history of HIV, HBV, HCV
* drug addiction
* vaccination within 4 weeks prior to study or planned vaccination during study
* prior receipt of any Zika vaccine
* recent infection 1 week prior to screening
* relevant medical history interfering with aim of study
* neoplastic disease, hematological malignancy
* history of autoimmune disease
* psychological condition that affects ability to participate in the study
* history of severe adverse reactions to vaccine administration
* history of anaphylaxis
* allergic reactions, abnormal lab values, or concomitant medication per decision of the investigator
* use of immunosuppressive drugs within 30 days before screening or planned use during study
* receipt of blood products within 120 days before screening or planned use during study
* pregnancy, unreliable contraception method
* decision of the investigator
* regular blood plasma donor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: Functional anti-Zika antibodies as measured by PRNT | 56 days
  Functional anti-Zika antibodies as measured by PRNT.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Austria (2):
  - Medical University of Vienna, Center for Pathophysiology, Infectiology and Immunology, Vienna
  - Medical University of Vienna, Department of Clinical Pharmacology, Vienna

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php